CLINICAL TRIAL: NCT06182475
Title: Increasing Equity in Live Donor Kidney Transplantation Through Effective Patient-Provider Communication
Brief Title: Development and Test of a Communication Skills Training for Transplant Providers - Aims 2 & 3
Acronym: EPPComm
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Cooperman Barnabas Medical Center (Unknown)
Responsible Party: Principal Investigator, Heather Gardiner (Traino), Professor, Temple University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: R01DK134630 (NIH)
Record Dates: First submitted 2023-08-18; First posted 2023-12-27 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-04

CONDITIONS: Kidney Disease, Chronic; End Stage Renal Disease; Kidney Replacement
Keywords: Patient-Provider Communication; Live Donor Kideny Transplantation; Provider Training; Communication Skills Training
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: To provide preliminary data on the efficacy and acceptability of the training program, we will employ a pre-post study design, with providers serving as their own controls (Aim 2). We will then test the indirect effects of the training on providers' communication with patients, patient and provider factors and live donor kidney transplant process outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EPPCom Provider Training (Experimental): A highly engaging and interactive 60-minute, in-person communication skills training program will be developed as part of this project. Participating transplant providers will complete a brief online survey before (pre) and after (post) participating in the training.
  Interventions: Behavioral: EPPComm Provider Training

INTERVENTIONS:
Behavioral: EPPComm Provider Training — A curriculum will be developed to educate patients about LDKT and promote the search of potential living donors while supporting patients' values and cultural preferences. The curriculum will consist of two components: didactic education and skills-based communication. The didactic component provides evidence of the impact of patient-provider communication and LDKT process outcomes for Black and Caucasian patients. The skills-based component will build communication confidence leading discussions about LDKT. It provides instructions for the key communication skills needed to confidently assuage patients' concerns about LDKT/live donation and motivates patients to search for living donor. The following will be covered: providing LDKT information/answering questions, highlighting LDKT benefits, refuting live donation misinformation, and encouraging patients to seek living donors.

SUMMARY:
The goal of this clinical trial is to understand the communication occurring between Black and Caucasian patients and their transplant providers during transplant evaluation consultations and assess relationships between these communicative elements and patient and provider factors, patient-reported outcomes and living donor transplant outcomes - living donor referrals, evaluations, and transplants. We will use these findings to inform the development of a communication skills training for transplant providers and test the impact of the training on providers' communication about live donor kidney transplants with Black and Caucasian patients and living donor transplant outcomes.

The main questions it aims to answer are:

* How does the use of the use of instrumental, relational and affective communication by patients and providers during the transplant consultation differ by patient and provider factors, patient-reported outcomes and patient ethnicity?
* What elements of instrumental, relational and affective communication will be predictive of live donor kidney transplant (LDKT) process outcomes (LD inquiries and evaluations, and actual LDKTs)?

Participants will be asked to complete brief surveys before and after the transplant consultation and to give permission for the consultation to be audiorecorded.

This data will be used to develop a training to educate providers on the key communication factors predictive of LDKT process outcomes specific to Black and Caucasian patients, and provide guidance on their application during patient consultations. Researchers will then compare communication and patient-reported and LDKT process outcomes between trained and untrained providers to see whether the training has any effect on living donor inquiries and evaluations, and actual LDKTs.

DETAILED DESCRIPTION:
Live donor kidney transplant (LDKT) is the preferred treatment modality for patients with chronic and end-stage kidney disease. LDKT is less expensive than prolonged dialysis and offers improved mortality and morbidity over either dialysis or deceased donor kidney transplants (DDKT). However, ethnic minorities have significantly less access to LDKT than their White counterparts. Collectively, Blacks, Asians, and Hispanics represent 64.3% of the kidney transplant wait list, yet received only 36% of all LDKTs in 2019. Further, rates of LDKTs have decreased for Black patients over the last decade. Decades of research point to patient-provider communication as a contributing factor to observed disparities in health and healthcare outcomes. To date, however, no attempt has been made to gauge the impact of the communication occurring during transplant evaluation consultations on LDKT outcomes. The long-term goal of the proposed study entitled, Increasing Equity in Live Donor Kidney Transplant through Effective Patient-Provider Communication, is to increase parity in access to LDKT for Black patients. A community-engaged, mixed-methods study employing a concurrent triangulation design is proposed to identify the specific communicative behaviors that result in live donor inquiries and evaluations, and actual LDKTs for Caucasian and Black patients, providing critical information to the design of an intervention to improve patient-provider communication about LDKT. Specifically, this project will simultaneously quantitatively assess patient and provider factors with established and hypothesized associations with receipt of LDKTs, and qualitatively assess discrete elements of patient-provider communication occurring during transplant evaluation consultations for Caucasian and Black patients (Aim 1). Brief quantitative surveys administered before and after medical consultations held as part of the evaluation for transplant candidacy will capture providers' (N=52) confidence and comfort discussing LDKT and patients' satisfaction with the consultation, medical mistrust, health literacy, and LDKT knowledge, attitudes and readiness. In addition, transplant evaluation consultations will be evaluated for 60 Caucasian and 60 Black patients (N=120) across the two study sites - Saint Barnabas Medical Center (NJ) and Temple University Hospital (PA), and qualitatively assess the communication occurring during the consultations. The findings will be used to inform development of the content and format of a communication skills training for transplant providers and evaluate the direct and indirect effects of the training on patient-reported and LDKT process outcomes (Aims 2 & 3). Intervening at the provider level is both practical, given that all transplant candidates already must undergo this consultation, and efficient, given that a single transplant physician can evaluate >100 transplant candidates per year. Thus, the results of this innovative study have the potential to increase access to LDKT for Black patients currently awaiting kidney transplant. Improving communication during the transplant consultation may prove to be an effective and efficient means of alleviating ethnic disparities in LDKT.

ELIGIBILITY:
Inclusion Criteria:

* (1) appear for a kidney transplant evaluation at Cooperman Barnabas Medical Center (CBMC) or Temple University Hospital (TUH)
* (2) speak English
* (3) be of self-reported Black or Caucasian ethnicity
* (4) be ≥18 years of age.

Including patients who:

1. have received prior kidney transplants
2. patients with limited English proficiency, as long as they speak with the physician via a translator
3. patients evaluated at offsite satellite locations that are not actually at CBMC or TUHS.

All transplant nephrologists, nurses, and social workers employed at the kidney transplant programs at CBMC and TUH who are actively involved in patient evaluations for transplant will be eligible for participation in the study. Providers refusing to permit digital audio recording of the transplant consultation will be deemed ineligible.

Exclusion Criteria:

* (1) are non-verbal or otherwise unable to converse with providers
* (2) are already listed for kidney transplant at CBMC or TUHS or at another transplant center
* (3) have limited English proficiency and speak directly with the physician in a language other than English.

Patients having (1) received an offer to donate a kidney from a family member or friend, or (2) explicitly asked a family member or friend to consider serving as a LD will be excluded, along with any patients refusing to permit digital audio recording of the transplant consultation will also be deemed ineligible to participate.

The following special populations will be excluded: adults unable to consent, individuals who are not yet adults (infants, children, teenagers), prisoners, and individuals who do not understand English.

It is unlikely that any female patient will be pregnant while awaiting kidney transplant; however, we will not exclude pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Live donor inquiries | Through study completion, 4 years
  Whether potential donors return a completed donor referral form to the patient's transplant program (yes/no)
Live donor evaluations | Through study completion, 4 years
  Whether potential donor appears, in-person, for the donor evaluation (yes/no)
Live donor kidney transplant | Through study completion, 4 years
  Whether patient receives a live donor kidney transplant (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Francis Weng, MD, Principal Investigator — St. Barnabas Medical Center
Locations (2):
- United States (2):
  - Cooperman Barnabas Medical Center, Livingston, New Jersey
  - Temple University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] United States Renal Data System. 2020 USRDS annual data report: Epidemiology of kidney disease in the United States. Executive Summary. National Institutes of Health, National Institute of Diabetes and Digestive and Kidney Diseases, Bethesda, MD, 2020. https://adr.usrds.org/2020. Accessed February 1, 2022.
- [Background] Haller MC, Kammer M, Oberbauer R. Dialysis vintage and outcomes in renal transplantation. Nephrol Dial Transplant. 2019 Apr 1;34(4):555-560. doi: 10.1093/ndt/gfy099. PMID 29897595
- [Background] Kaballo MA, Canney M, O'Kelly P, Williams Y, O'Seaghdha CM, Conlon PJ. A comparative analysis of survival of patients on dialysis and after kidney transplantation. Clin Kidney J. 2018 Jun;11(3):389-393. doi: 10.1093/ckj/sfx117. Epub 2017 Oct 18. PMID 29942504
- [Background] Wyld M, Morton RL, Hayen A, Howard K, Webster AC. A systematic review and meta-analysis of utility-based quality of life in chronic kidney disease treatments. PLoS Med. 2012;9(9):e1001307. doi: 10.1371/journal.pmed.1001307. Epub 2012 Sep 11. PMID 22984353
- [Background] Organ Procurement and Transplantation Network. U.S. Department of Health and Human Services. https://optn.transplant.hrsa.gov/data/view-data-reports/national-data/#. Accessed February 1, 2022.
- [Background] United States Renal Data System. 2018 USRDS annual data report: Epidemiology of kidney disease in the United States. National Institutes of Health, National Institute of Diabetes and Digestive and Kidney Diseases, Bethesda, MD, 2018. https://www.usrds.org/2018/view/Default.aspx. Accessed February 1, 2022.
- [Background] Navaneethan SD, Singh S. A systematic review of barriers in access to renal transplantation among African Americans in the United States. Clin Transplant. 2006 Nov-Dec;20(6):769-75. doi: 10.1111/j.1399-0012.2006.00568.x. PMID 17100728
- [Background] Waterman AD, Peipert JD, Xiao H, Goalby CJ, Kawakita S, Cui Y, Lentine KL. Education Strategies in Dialysis Centers Associated With Increased Transplant Wait-listing Rates. Transplantation. 2020 Feb;104(2):335-342. doi: 10.1097/TP.0000000000002781. PMID 31335777
- [Background] Kutner NG, Zhang R, Huang Y, Johansen KL. Impact of race on predialysis discussions and kidney transplant preemptive wait-listing. Am J Nephrol. 2012;35(4):305-11. doi: 10.1159/000336891. Epub 2012 Mar 9. PMID 22414927
- [Background] Browne T, Patzer RE, Gander J, Amamoo MA, Krisher J, Sauls L, Pastan S. Kidney transplant referral practices in southeastern dialysis units. Clin Transplant. 2016 Apr;30(4):365-71. doi: 10.1111/ctr.12693. Epub 2016 Feb 12. PMID 26782140
- [Background] Jones D, You Z, Kendrick JB. Racial/Ethnic Differences in Barriers to Kidney Transplant Evaluation among Hemodialysis Patients. Am J Nephrol. 2018;47(1):1-7. doi: 10.1159/000484484. Epub 2017 Dec 19. PMID 29258094
- [Background] Nonterah CW, Gardiner HM. Pre-transplant evaluation completion for Black/African American renal patients: Two theoretical frameworks. Patient Educ Couns. 2020 May;103(5):988-998. doi: 10.1016/j.pec.2019.11.005. Epub 2019 Nov 9. PMID 31733984
- [Background] Taber DJ, Gebregziabher M, Hunt KJ, Srinivas T, Chavin KD, Baliga PK, Egede LE. Twenty years of evolving trends in racial disparities for adult kidney transplant recipients. Kidney Int. 2016 Oct;90(4):878-87. doi: 10.1016/j.kint.2016.06.029. Epub 2016 Aug 20. PMID 27555121
- [Background] Ng YH, Pankratz VS, Leyva Y, Ford CG, Pleis JR, Kendall K, Croswell E, Dew MA, Shapiro R, Switzer GE, Unruh ML, Myaskovsky L. Does Racial Disparity in Kidney Transplant Waitlisting Persist After Accounting for Social Determinants of Health? Transplantation. 2020 Jul;104(7):1445-1455. doi: 10.1097/TP.0000000000003002. PMID 31651719
- [Background] Friedewald JJ, Samana CJ, Kasiske BL, Israni AK, Stewart D, Cherikh W, Formica RN. The kidney allocation system. Surg Clin North Am. 2013 Dec;93(6):1395-406. doi: 10.1016/j.suc.2013.08.007. PMID 24206858
- [Background] Kulkarni S, Ladin K, Haakinson D, Greene E, Li L, Deng Y. Association of Racial Disparities With Access to Kidney Transplant After the Implementation of the New Kidney Allocation System. JAMA Surg. 2019 Jul 1;154(7):618-625. doi: 10.1001/jamasurg.2019.0512. PMID 30942882
- [Background] Martins PN, Mustian MN, MacLennan PA, Ortiz JA, Akoad M, Caicedo JC, Echeverri GJ, Gray SH, Lopez-Soler RI, Gunasekaran G, Kelly B, Mobley CM, Black SM, Esquivel C, Locke JE. Impact of the new kidney allocation system A2/A2B --> B policy on access to transplantation among minority candidates. Am J Transplant. 2018 Aug;18(8):1947-1953. doi: 10.1111/ajt.14719. Epub 2018 Mar 31. PMID 29509285
- [Background] Wilkins LJ, Nyame YA, Gan V, Lin S, Greene DJ, Flechner SM, Modlin CS. A Contemporary Analysis of Outcomes and Modifiable Risk Factors of Ethnic Disparities in Kidney Transplantation. J Natl Med Assoc. 2019 Apr;111(2):202-209. doi: 10.1016/j.jnma.2018.10.011. Epub 2018 Nov 6. PMID 30409716
- [Background] Purnell TS, Luo X, Cooper LA, Massie AB, Kucirka LM, Henderson ML, Gordon EJ, Crews DC, Boulware LE, Segev DL. Association of Race and Ethnicity With Live Donor Kidney Transplantation in the United States From 1995 to 2014. JAMA. 2018 Jan 2;319(1):49-61. doi: 10.1001/jama.2017.19152. PMID 29297077
- [Background] Joshi S, Gaynor JJ, Bayers S, Guerra G, Eldefrawy A, Chediak Z, Companioni L, Sageshima J, Chen L, Kupin W, Roth D, Mattiazzi A, Burke GW 3rd, Ciancio G. Disparities among Blacks, Hispanics, and Whites in time from starting dialysis to kidney transplant waitlisting. Transplantation. 2013 Jan 27;95(2):309-18. doi: 10.1097/TP.0b013e31827191d4. PMID 23325005
- [Background] Rodrigue JR, Paek MJ, Egbuna O, Waterman AD, Schold JD, Pavlakis M, Mandelbrot DA. Readiness of wait-listed black patients to pursue live donor kidney transplant. Prog Transplant. 2014 Dec;24(4):355-61. doi: 10.7182/pit2014337. PMID 25488559
- [Background] Purnell TS, Hall YN, Boulware LE. Understanding and overcoming barriers to living kidney donation among racial and ethnic minorities in the United States. Adv Chronic Kidney Dis. 2012 Jul;19(4):244-51. doi: 10.1053/j.ackd.2012.01.008. PMID 22732044
- [Background] Waterman AD, Rodrigue JR, Purnell TS, Ladin K, Boulware LE. Addressing racial and ethnic disparities in live donor kidney transplantation: priorities for research and intervention. Semin Nephrol. 2010 Jan;30(1):90-8. doi: 10.1016/j.semnephrol.2009.10.010. PMID 20116653
- [Background] Rodrigue JR, Kazley AS, Mandelbrot DA, Hays R, LaPointe Rudow D, Baliga P; American Society of Transplantation. Living Donor Kidney Transplantation: Overcoming Disparities in Live Kidney Donation in the US--Recommendations from a Consensus Conference. Clin J Am Soc Nephrol. 2015 Sep 4;10(9):1687-95. doi: 10.2215/CJN.00700115. Epub 2015 Apr 16. PMID 25883072
- [Background] Harding K, Mersha TB, Pham PT, Waterman AD, Webb FA, Vassalotti JA, Nicholas SB. Health Disparities in Kidney Transplantation for African Americans. Am J Nephrol. 2017;46(2):165-175. doi: 10.1159/000479480. Epub 2017 Aug 5. PMID 28787713
- [Background] Sieverdes JC, Nemeth LS, Magwood GS, Baliga PK, Chavin KD, Ruggiero KJ, Treiber FA. African American kidney transplant patients' perspectives on challenges in the living donation process. Prog Transplant. 2015 Jun;25(2):164-75. doi: 10.7182/pit2015852. PMID 26107278
- [Background] Waterman AD, Peipert JD, Hyland SS, McCabe MS, Schenk EA, Liu J. Modifiable patient characteristics and racial disparities in evaluation completion and living donor transplant. Clin J Am Soc Nephrol. 2013 Jun;8(6):995-1002. doi: 10.2215/CJN.08880812. Epub 2013 Mar 21. PMID 23520044
- [Background] Davis LA, Grogan TM, Cox J, Weng FL. Inter- and Intrapersonal Barriers to Living Donor Kidney Transplant among Black Recipients and Donors. J Racial Ethn Health Disparities. 2017 Aug;4(4):671-679. doi: 10.1007/s40615-016-0270-8. Epub 2016 Aug 12. PMID 27519479
- [Background] Weng FL, Reese PP, Mulgaonkar S, Patel AM. Barriers to living donor kidney transplantation among black or older transplant candidates. Clin J Am Soc Nephrol. 2010 Dec;5(12):2338-47. doi: 10.2215/CJN.03040410. Epub 2010 Sep 28. PMID 20876682
- [Background] Weng FL, Dhillon N, Lin Y, Mulgaonkar S, Patel AM. Racial differences in outcomes of the evaluation of potential live kidney donors: a retrospective cohort study. Am J Nephrol. 2012;35(5):409-15. doi: 10.1159/000337949. Epub 2012 Apr 19. PMID 22517188
- [Background] Norman SP, Song PX, Hu Y, Ojo AO. Transition from donor candidates to live kidney donors: the impact of race and undiagnosed medical disease states. Clin Transplant. 2011 Jan-Feb;25(1):136-45. doi: 10.1111/j.1399-0012.2009.01188.x. PMID 20047616
- [Background] Lunsford SL, Simpson KS, Chavin KD, Menching KJ, Miles LG, Shilling LM, Smalls GR, Baliga PK. Racial disparities in living kidney donation: is there a lack of willing donors or an excess of medically unsuitable candidates? Transplantation. 2006 Oct 15;82(7):876-81. doi: 10.1097/01.tp.0000232693.69773.42. PMID 17038900
- [Background] Traino HM. Communication self-efficacy, perceived conversational difficulty, and renal patients' discussions about transplantation. Patient Educ Couns. 2014 Feb;94(2):180-6. doi: 10.1016/j.pec.2013.10.012. Epub 2013 Nov 5. PMID 24280037
- [Background] Waterman AD, Barrett AC, Stanley SL. Optimal transplant education for recipients to increase pursuit of living donation. Prog Transplant. 2008 Mar;18(1):55-62. doi: 10.1177/152692480801800111. PMID 18429583
- [Background] Boulware LE, Meoni LA, Fink NE, Parekh RS, Kao WH, Klag MJ, Powe NR. Preferences, knowledge, communication and patient-physician discussion of living kidney transplantation in African American families. Am J Transplant. 2005 Jun;5(6):1503-12. doi: 10.1111/j.1600-6143.2005.00860.x. PMID 15888061
- [Background] DePasquale N, Ellis MJ, Sudan DL, Ephraim PL, McElroy LM, Mohottige D, Davenport CA, Zhang X, Peskoe SB, Strigo TS, Cabacungan AN, Pounds I, Riley JA, Falkovic M, Boulware LE. African Americans' discussions about living-donor kidney transplants with family or friends: Who, what, and why not? Clin Transplant. 2021 Apr;35(4):e14222. doi: 10.1111/ctr.14222. Epub 2021 Jan 25. PMID 33423353
- [Background] Arriola KR, Powell CL, Thompson NJ, Perryman JP, Basu M. Living donor transplant education for African American patients with end-stage renal disease. Prog Transplant. 2014 Dec;24(4):362-70. doi: 10.7182/pit2014830. PMID 25488560
- [Background] Boulware LE, Hill-Briggs F, Kraus ES, Melancon JK, Falcone B, Ephraim PL, Jaar BG, Gimenez L, Choi M, Senga M, Kolotos M, Lewis-Boyer L, Cook C, Light L, DePasquale N, Noletto T, Powe NR. Effectiveness of educational and social worker interventions to activate patients' discussion and pursuit of preemptive living donor kidney transplantation: a randomized controlled trial. Am J Kidney Dis. 2013 Mar;61(3):476-86. doi: 10.1053/j.ajkd.2012.08.039. Epub 2012 Oct 22. PMID 23089512
- [Background] Weng FL, Brown DR, Peipert JD, Holland B, Waterman AD. Protocol of a cluster randomized trial of an educational intervention to increase knowledge of living donor kidney transplant among potential transplant candidates. BMC Nephrol. 2013 Nov 19;14:256. doi: 10.1186/1471-2369-14-256. PMID 24245948
- [Background] Waterman AD, McSorley AM, Peipert JD, Goalby CJ, Peace LJ, Lutz PA, Thein JL. Explore Transplant at Home: a randomized control trial of an educational intervention to increase transplant knowledge for Black and White socioeconomically disadvantaged dialysis patients. BMC Nephrol. 2015 Aug 28;16:150. doi: 10.1186/s12882-015-0143-0. PMID 26316264
- [Background] Gordon EJ, Feinglass J, Carney P, Vera K, Olivero M, Black A, O'Connor KG, Baumgart JM, Caicedo JC. A Website Intervention to Increase Knowledge About Living Kidney Donation and Transplantation Among Hispanic/Latino Dialysis Patients. Prog Transplant. 2016 Mar;26(1):82-91. doi: 10.1177/1526924816632124. PMID 27136254
- [Background] Gordon EJ, Feinglass J, Carney P, Vera K, Olivero M, Black A, O'Connor K, MacLean J, Nichols S, Sageshima J, Preczewski L, Caicedo JC. A Culturally Targeted Website for Hispanics/Latinos About Living Kidney Donation and Transplantation: A Randomized Controlled Trial of Increased Knowledge. Transplantation. 2016 May;100(5):1149-60. doi: 10.1097/TP.0000000000000932. PMID 26444846
- [Background] Traino HM, West SM, Nonterah CW, Russell J, Yuen E. Communicating About Choices in Transplantation (COACH). Prog Transplant. 2017 Mar;27(1):31-38. doi: 10.1177/1526924816679844. Epub 2016 Nov 25. PMID 27888276
- [Background] Rodrigue JR, Cornell DL, Lin JK, Kaplan B, Howard RJ. Increasing live donor kidney transplantation: a randomized controlled trial of a home-based educational intervention. Am J Transplant. 2007 Feb;7(2):394-401. doi: 10.1111/j.1600-6143.2006.01623.x. Epub 2006 Dec 6. PMID 17173659
- [Background] Pradel FG, Suwannaprom P, Mullins CD, Sadler J, Bartlett ST. Short-term impact of an educational program promoting live donor kidney transplantation in dialysis centers. Prog Transplant. 2008 Dec;18(4):263-72. doi: 10.1177/152692480801800409. PMID 19186579
- [Background] Rodrigue JR, Paek MJ, Egbuna O, Waterman AD, Schold JD, Pavlakis M, Mandelbrot DA. Making house calls increases living donor inquiries and evaluations for blacks on the kidney transplant waiting list. Transplantation. 2014 Nov 15;98(9):979-86. doi: 10.1097/TP.0000000000000165. PMID 24825528
- [Background] Waterman AD, Robbins ML, Paiva AL, Peipert JD, Kynard-Amerson CS, Goalby CJ, Davis LA, Thein JL, Schenk EA, Baldwin KA, Skelton SL, Amoyal NR, Brick LA. Your Path to Transplant: a randomized controlled trial of a tailored computer education intervention to increase living donor kidney transplant. BMC Nephrol. 2014 Oct 14;15:166. doi: 10.1186/1471-2369-15-166. PMID 25315644
- [Background] Waterman AD, Peipert JD, McSorley AM, Goalby CJ, Beaumont JL, Peace L. Direct Delivery of Kidney Transplant Education to Black and Low-Income Patients Receiving Dialysis: A Randomized Controlled Trial. Am J Kidney Dis. 2019 Nov;74(5):640-649. doi: 10.1053/j.ajkd.2019.03.430. Epub 2019 Jun 19. PMID 31227225
- [Background] Strigo TS, Ephraim PL, Pounds I, Hill-Briggs F, Darrell L, Ellis M, Sudan D, Rabb H, Segev D, Wang NY, Kaiser M, Falkovic M, Lebov JF, Boulware LE. The TALKS study to improve communication, logistical, and financial barriers to live donor kidney transplantation in African Americans: protocol of a randomized clinical trial. BMC Nephrol. 2015 Oct 9;16:160. doi: 10.1186/s12882-015-0153-y. PMID 26452366
- [Background] Kumar K, King EA, Muzaale AD, Konel JM, Bramstedt KA, Massie AB, Segev DL, Cameron AM. A Smartphone App for Increasing Live Organ Donation. Am J Transplant. 2016 Dec;16(12):3548-3553. doi: 10.1111/ajt.13961. Epub 2016 Aug 10. PMID 27402293
- [Background] Garonzik-Wang JM, Berger JC, Ros RL, Kucirka LM, Deshpande NA, Boyarsky BJ, Montgomery RA, Hall EC, James NT, Segev DL. Live donor champion: finding live kidney donors by separating the advocate from the patient. Transplantation. 2012 Jun 15;93(11):1147-50. doi: 10.1097/TP.0b013e31824e75a5. PMID 22461037
- [Background] Moore DR, Feurer ID, Zavala EY, Shaffer D, Karp S, Hoy H, Moore DE. A web-based application for initial screening of living kidney donors: development, implementation and evaluation. Am J Transplant. 2013 Feb;13(2):450-7. doi: 10.1111/j.1600-6143.2012.04340.x. Epub 2012 Dec 3. PMID 23205926
- [Background] Rodrigue JR, Cornell DL, Kaplan B, Howard RJ. A randomized trial of a home-based educational approach to increase live donor kidney transplantation: effects in blacks and whites. Am J Kidney Dis. 2008 Apr;51(4):663-70. doi: 10.1053/j.ajkd.2007.11.027. Epub 2008 Mar 4. PMID 18371542
- [Background] Ismail SY, Luchtenburg AE, Timman R, Zuidema WC, Boonstra C, Weimar W, Busschbach JJ, Massey EK. Home-based family intervention increases knowledge, communication and living donation rates: a randomized controlled trial. Am J Transplant. 2014 Aug;14(8):1862-9. doi: 10.1111/ajt.12751. Epub 2014 Jun 16. PMID 24935081
- [Background] Taber DJ, Gebregziabher M, Srinivas T, Egede LE, Baliga PK. Transplant Center Variability in Disparities for African-American Kidney Transplant Recipients. Ann Transplant. 2018 Feb 16;23:119-128. doi: 10.12659/aot.907226. PMID 29449524
- [Background] Hall EC, James NT, Garonzik Wang JM, Berger JC, Montgomery RA, Dagher NN, Desai NM, Segev DL. Center-level factors and racial disparities in living donor kidney transplantation. Am J Kidney Dis. 2012 Jun;59(6):849-57. doi: 10.1053/j.ajkd.2011.12.021. Epub 2012 Feb 25. PMID 22370021
- [Background] Hunt HF, Rodrigue JR, Dew MA, Schaffer RL, Henderson ML, Bloom R, Kacani P, Shim P, Bolton L, Sanchez W, Lentine KL. Strategies for Increasing Knowledge, Communication, and Access to Living Donor Transplantation: an Evidence Review to Inform Patient Education. Curr Transplant Rep. 2018 Mar;5(1):27-44. doi: 10.1007/s40472-018-0181-1. Epub 2018 Feb 5. PMID 30873335
- [Background] Sandal S, Charlebois K, Fiore JF Jr, Wright DK, Fortin MC, Feldman LS, Alam A, Weber C. Health Professional-Identified Barriers to Living Donor Kidney Transplantation: A Qualitative Study. Can J Kidney Health Dis. 2019 Feb 13;6:2054358119828389. doi: 10.1177/2054358119828389. eCollection 2019. PMID 30792874
- [Background] Paskett E, Thompson B, Ammerman AS, Ortega AN, Marsteller J, Richardson D. Multilevel Interventions To Address Health Disparities Show Promise In Improving Population Health. Health Aff (Millwood). 2016 Aug 1;35(8):1429-34. doi: 10.1377/hlthaff.2015.1360. PMID 27503968
- [Background] Gorin SS, Badr H, Krebs P, Prabhu Das I. Multilevel interventions and racial/ethnic health disparities. J Natl Cancer Inst Monogr. 2012 May;2012(44):100-11. doi: 10.1093/jncimonographs/lgs015. PMID 22623602
- [Background] Thomas SB, Quinn SC, Butler J, Fryer CS, Garza MA. Toward a fourth generation of disparities research to achieve health equity. Annu Rev Public Health. 2011;32:399-416. doi: 10.1146/annurev-publhealth-031210-101136. PMID 21219164
- [Background] Weng FL, Peipert JD, Holland BK, Brown DR, Waterman AD. A Clustered Randomized Trial of an Educational Intervention During Transplant Evaluation to Increase Knowledge of Living Donor Kidney Transplant. Prog Transplant. 2017 Dec;27(4):377-385. doi: 10.1177/1526924817732021. Epub 2017 Sep 19. PMID 29187135
- [Background] Ong LM, de Haes JC, Hoos AM, Lammes FB. Doctor-patient communication: a review of the literature. Soc Sci Med. 1995 Apr;40(7):903-18. doi: 10.1016/0277-9536(94)00155-m. PMID 7792630
- [Background] Stewart MA. Effective physician-patient communication and health outcomes: a review. CMAJ. 1995 May 1;152(9):1423-33. PMID 7728691
- [Background] Riedl D, Schussler G. The Influence of Doctor-Patient Communication on Health Outcomes: A Systematic Review. Z Psychosom Med Psychother. 2017 Jun;63(2):131-150. doi: 10.13109/zptm.2017.63.2.131. No abstract available. PMID 28585507
- [Background] Henry SG, Fuhrel-Forbis A, Rogers MA, Eggly S. Association between nonverbal communication during clinical interactions and outcomes: a systematic review and meta-analysis. Patient Educ Couns. 2012 Mar;86(3):297-315. doi: 10.1016/j.pec.2011.07.006. Epub 2011 Aug 6. PMID 21824738
- [Background] Lafata JE, Cooper G, Divine G, Oja-Tebbe N, Flocke SA. Patient-physician colorectal cancer screening discussion content and patients' use of colorectal cancer screening. Patient Educ Couns. 2014 Jan;94(1):76-82. doi: 10.1016/j.pec.2013.09.008. Epub 2013 Sep 17. PMID 24094919
- [Background] Mosen DM, Feldstein AC, Perrin NA, Rosales AG, Smith DH, Liles EG, Schneider JL, Meyers RE, Elston-Lafata J. More comprehensive discussion of CRC screening associated with higher screening. Am J Manag Care. 2013 Apr;19(4):265-71. PMID 23725359
- [Background] Siminoff LA, Traino HM, Gordon NH. An exploratory study of relational, persuasive, and nonverbal communication in requests for tissue donation. J Health Commun. 2011 Oct;16(9):955-75. doi: 10.1080/10810730.2011.561908. Epub 2011 May 24. PMID 21512935
- [Background] Traino HM, Siminoff LA. Keep it going: maintaining health conversations using relational and instrumental approaches. Health Commun. 2016;31(3):308-19. doi: 10.1080/10410236.2014.950020. Epub 2015 Sep 1. PMID 26325602
- [Background] Dorflinger L, Auerbach SM, Siminoff LA. Predictors of consent in tissue donation: interpersonal aspects and information provision during requests by phone. Patient Educ Couns. 2013 May;91(2):161-6. doi: 10.1016/j.pec.2012.12.003. Epub 2012 Dec 28. PMID 23276387
- [Background] Kaplan SH, Greenfield S, Ware JE Jr. Assessing the effects of physician-patient interactions on the outcomes of chronic disease. Med Care. 1989 Mar;27(3 Suppl):S110-27. doi: 10.1097/00005650-198903001-00010. PMID 2646486
- [Background] Beck RS, Daughtridge R, Sloane PD. Physician-patient communication in the primary care office: a systematic review. J Am Board Fam Pract. 2002 Jan-Feb;15(1):25-38. PMID 11841136
- [Background] Chawla N, Blanch-Hartigan D, Virgo KS, Ekwueme DU, Han X, Forsythe L, Rodriguez J, McNeel TS, Yabroff KR. Quality of Patient-Provider Communication Among Cancer Survivors: Findings From a Nationally Representative Sample. J Oncol Pract. 2016 Dec;12(12):e964-e973. doi: 10.1200/JOP.2015.006999. Epub 2016 Oct 31. PMID 27221992
- [Background] Tongue JR, Epps HR, Forese LL. Communication skills for patient-centered care: research-based, easily learned techniques for medical interviews that benefit orthopaedic surgeons and their patients. J Bone Joint Surg Am. 2005;87:652-58. PMID:
- [Background] Bao Y, Fox SA, Escarce JJ. Socioeconomic and racial/ethnic differences in the discussion of cancer screening: "between-" versus "within-" physician differences. Health Serv Res. 2007 Jun;42(3 Pt 1):950-70. doi: 10.1111/j.1475-6773.2006.00638.x. PMID 17489898
- [Background] Palmer NR, Kent EE, Forsythe LP, Arora NK, Rowland JH, Aziz NM, Blanch-Hartigan D, Oakley-Girvan I, Hamilton AS, Weaver KE. Racial and ethnic disparities in patient-provider communication, quality-of-care ratings, and patient activation among long-term cancer survivors. J Clin Oncol. 2014 Dec 20;32(36):4087-94. doi: 10.1200/JCO.2014.55.5060. Epub 2014 Nov 17. PMID 25403220
- [Background] Trenchard L, Mc Grath-Lone L, Ward H. Ethnic variation in cancer patients' ratings of information provision, communication and overall care. Ethn Health. 2016 Oct;21(5):515-33. doi: 10.1080/13557858.2015.1126561. Epub 2016 Feb 7. PMID 26853061
- [Background] Johnson RL, Roter D, Powe NR, Cooper LA. Patient race/ethnicity and quality of patient-physician communication during medical visits. Am J Public Health. 2004 Dec;94(12):2084-90. doi: 10.2105/ajph.94.12.2084. PMID 15569958
- [Background] Martin KD, Roter DL, Beach MC, Carson KA, Cooper LA. Physician communication behaviors and trust among black and white patients with hypertension. Med Care. 2013 Feb;51(2):151-7. doi: 10.1097/MLR.0b013e31827632a2. PMID 23132201
- [Background] Beach MC, Saha S, Korthuis PT, Sharp V, Cohn J, Wilson IB, Eggly S, Cooper LA, Roter D, Sankar A, Moore R. Patient-provider communication differs for black compared to white HIV-infected patients. AIDS Behav. 2011 May;15(4):805-11. doi: 10.1007/s10461-009-9664-5. PMID 20066486
- [Background] Beach MC, Saha S, Korthuis PT, Sharp V, Cohn J, Wilson I, Eggly S, Cooper LA, Roter D, Sankar A, Moore R. Differences in patient-provider communication for Hispanic compared to non-Hispanic white patients in HIV care. J Gen Intern Med. 2010 Jul;25(7):682-7. doi: 10.1007/s11606-010-1310-4. Epub 2010 Mar 18. PMID 20238204
- [Background] Cene CW, Roter D, Carson KA, Miller ER 3rd, Cooper LA. The effect of patient race and blood pressure control on patient-physician communication. J Gen Intern Med. 2009 Sep;24(9):1057-64. doi: 10.1007/s11606-009-1051-4. Epub 2009 Jul 3. PMID 19575270
- [Background] Ghods BK, Roter DL, Ford DE, Larson S, Arbelaez JJ, Cooper LA. Patient-physician communication in the primary care visits of African Americans and whites with depression. J Gen Intern Med. 2008 May;23(5):600-6. doi: 10.1007/s11606-008-0539-7. Epub 2008 Feb 9. PMID 18264834
- [Background] Cooper-Patrick L, Gallo JJ, Gonzales JJ, Vu HT, Powe NR, Nelson C, Ford DE. Race, gender, and partnership in the patient-physician relationship. JAMA. 1999 Aug 11;282(6):583-9. doi: 10.1001/jama.282.6.583. PMID 10450723
- [Background] Balkrishnan R, Dugan E, Camacho FT, Hall MA. Trust and satisfaction with physicians, insurers, and the medical profession. Med Care. 2003 Sep;41(9):1058-64. doi: 10.1097/01.MLR.0000083743.15238.9F. PMID 12972845
- [Background] Cooper LA, Roter DL, Johnson RL, Ford DE, Steinwachs DM, Powe NR. Patient-centered communication, ratings of care, and concordance of patient and physician race. Ann Intern Med. 2003 Dec 2;139(11):907-15. doi: 10.7326/0003-4819-139-11-200312020-00009. PMID 14644893
- [Background] White RO, Chakkalakal RJ, Presley CA, Bian A, Schildcrout JS, Wallston KA, Barto S, Kripalani S, Rothman R. Perceptions of Provider Communication Among Vulnerable Patients With Diabetes: Influences of Medical Mistrust and Health Literacy. J Health Commun. 2016;21(sup2):127-134. doi: 10.1080/10810730.2016.1207116. Epub 2016 Sep 23. PMID 27662442
- [Background] Eveland WP. The effect of political discussion in producing informed citizens: The roles of information, motivation, and elaboration. Pol Commun. 2004;21:177-193.
- [Background] Southwell BG, Yzer MC. The roles of interpersonal communication in mass media campaigns. Ann Int Commun Assoc. 2007;31:420-262
- [Background] Tavakoly Sany SB, Behzhad F, Ferns G, Peyman N. Communication skills training for physicians improves health literacy and medical outcomes among patients with hypertension: a randomized controlled trial. BMC Health Serv Res. 2020 Jan 23;20(1):60. doi: 10.1186/s12913-020-4901-8. PMID 31973765
- [Background] Norgaard B, Kofoed PE, Ohm Kyvik K, Ammentorp J. Communication skills training for health care professionals improves the adult orthopaedic patient's experience of quality of care. Scand J Caring Sci. 2012 Dec;26(4):698-704. doi: 10.1111/j.1471-6712.2012.00982.x. Epub 2012 Mar 16. PMID 22420418
- [Background] Siminoff LA, Traino HM, Genderson MW. Communicating Effectively about Organ Donation: A Randomized Trial of a Behavioral Communication Intervention to Improve Discussions about Donation. Transplant Direct. 2015 Mar;1(2):e5. doi: 10.1097/TXD.0000000000000513. PMID 26146659
- [Background] Siminoff LA, Marshall HM, Dumenci L, Bowen G, Swaminathan A, Gordon N. Communicating effectively about donation: an educational intervention to increase consent to donation. Prog Transplant. 2009 Mar;19(1):35-43. doi: 10.1177/152692480901900105. PMID 19341061
- [Background] Siminoff LA, Gardiner HM, Alolod GP, Wilson-Genderson M. Using Online Communication Skills Training to Increase Organ Donation Authorization. Prog Transplant. 2020 Sep;30(3):212-219. doi: 10.1177/1526924820933846. PMID 32783529
- [Background] Trickey AW, Newcomb AB, Porrey M, Piscitani F, Wright J, Graling P, Dort J. Two-Year Experience Implementing a Curriculum to Improve Residents' Patient-Centered Communication Skills. J Surg Educ. 2017 Nov-Dec;74(6):e124-e132. doi: 10.1016/j.jsurg.2017.07.014. Epub 2017 Jul 26. PMID 28756146
- [Background] Berlacher K, Arnold RM, Reitschuler-Cross E, Teuteberg J, Teuteberg W. The Impact of Communication Skills Training on Cardiology Fellows' and Attending Physicians' Perceived Comfort with Difficult Conversations. J Palliat Med. 2017 Jul;20(7):767-769. doi: 10.1089/jpm.2016.0509. Epub 2017 Mar 1. PMID 28437212
- [Background] Norgaard B, Ammentorp J, Ohm Kyvik K, Kofoed PE. Communication skills training increases self-efficacy of health care professionals. J Contin Educ Health Prof. 2012 Spring;32(2):90-7. doi: 10.1002/chp.21131. PMID 22733636
- [Background] Schell JO, Green JA, Tulsky JA, Arnold RM. Communication skills training for dialysis decision-making and end-of-life care in nephrology. Clin J Am Soc Nephrol. 2013 Apr;8(4):675-80. doi: 10.2215/CJN.05220512. Epub 2012 Nov 8. PMID 23143502
- [Background] Schell JO, Cohen RA, Green JA, Rubio D, Childers JW, Claxton R, Jeong K, Arnold RM. NephroTalk: Evaluation of a Palliative Care Communication Curriculum for Nephrology Fellows. J Pain Symptom Manage. 2018 Nov;56(5):767-773.e2. doi: 10.1016/j.jpainsymman.2018.08.002. Epub 2018 Aug 14. PMID 30118758
- [Background] Barth J, Lannen P. Efficacy of communication skills training courses in oncology: a systematic review and meta-analysis. Ann Oncol. 2011 May;22(5):1030-1040. doi: 10.1093/annonc/mdq441. Epub 2010 Oct 25. PMID 20974653
- [Background] Selman LE, Brighton LJ, Hawkins A, McDonald C, O'Brien S, Robinson V, Khan SA, George R, Ramsenthaler C, Higginson IJ, Koffman J. The Effect of Communication Skills Training for Generalist Palliative Care Providers on Patient-Reported Outcomes and Clinician Behaviors: A Systematic Review and Meta-analysis. J Pain Symptom Manage. 2017 Sep;54(3):404-416.e5. doi: 10.1016/j.jpainsymman.2017.04.007. Epub 2017 Aug 1. PMID 28778560
- [Background] Mortsiefer A, Rotthoff T, Schmelzer R, Immecke J, Ortmanns B, in der Schmitten J, Altiner A, Karger A. Implementation of the interdisciplinary curriculum Teaching and Assessing Communicative Competence in the fourth academic year of medical studies (CoMeD). GMS Z Med Ausbild. 2012;29(1):Doc06. doi: 10.3205/zma000776. Epub 2012 Feb 15. PMID 22403591
- [Background] Accreditation Council for Graduate Medical Education (ACGME). Common Program Requirements. 2018. https://www.acgme.org/What-We-Do/Accreditation/Common-Program-Requirements. Accessed February 1, 2022.
- [Background] Association of American Medical Colleges (AAMC). https://www.aamc.org/what-we-do/mission-areas/medical-education/msop. Accessed February 1, 2022.
- [Background] Siminoff LA, Traino HM, Gordon N. Determinants of family consent to tissue donation. J Trauma. 2010 Oct;69(4):956-63. doi: 10.1097/TA.0b013e3181d8924b. PMID 20526212
- [Background] Siminoff LA, Traino HM. Consenting to donation: an examination of current practices in informed consent for tissue donation in the US. Cell Tissue Bank. 2013 Mar;14(1):85-95. doi: 10.1007/s10561-012-9303-7. Epub 2012 Mar 8. PMID 22395736
- [Background] Traino HM, Nonterah CW, Gupta G, Mincemoyer J. Living Kidney Donors' Information Needs and Preferences. Prog Transplant. 2016 Mar;26(1):47-54. doi: 10.1177/1526924816633943. PMID 27136249
- [Background] Alolod GP, Gardiner H, Agu C, Turner JL, Kelly PJ, Siminoff LA, Gordon EJ, Norden R, Daly TA, Benitez A, Hernandez I, Guinansaca N, Winther LR, Bergeron CD, Montalvo A, Gonzalez T. A Culturally Targeted eLearning Module on Organ Donation (Promotoras de Donacion): Design and Development. J Med Internet Res. 2020 Jan 13;22(1):e15793. doi: 10.2196/15793. PMID 31929102
- [Background] Gillespie A, Hammer H, Lee J, Nnewihe C, Gordon J, Silva P. Lack of listing status awareness: results of a single-center survey of hemodialysis patients. Am J Transplant. 2011 Jul;11(7):1522-6. doi: 10.1111/j.1600-6143.2011.03524.x. Epub 2011 Apr 12. PMID 21486390
- [Background] Gillespie A, Hammer H, Kolenikov S, Polychronopoulou A, Ouzienko V, Obradovic Z, Urbanski MA, Browne T, Silva P. Sex differences and attitudes toward living donor kidney transplantation among urban black patients on hemodialysis. Clin J Am Soc Nephrol. 2014 Oct 7;9(10):1764-72. doi: 10.2215/CJN.12531213. Epub 2014 Aug 14. PMID 25125384
- [Background] Bauerle Bass S, Hollin IL, Kelly PJ, Alhajji M, D'Avanzo P, Maurer L, Gillespie A, Schatell D, Gardiner HM. Perceptions of live donor kidney transplantation: Use of segmentation analysis and perceptual mapping to understand differences by self-reported health status in people on dialysis. BMC Nephrology. In press
- [Background] Gillespie A, Gardiner HM, Fink EL, Reese PP, Gadegbeku CA, Obradovic Z. Does Sex, Race, and the Size of a Kidney Transplant Candidate's Social Network Affect the Number of Living Donor Requests? A Multicenter Social Network Analysis of Patients on the Kidney Transplant Waitlist. Transplantation. 2020 Dec;104(12):2632-2641. doi: 10.1097/TP.0000000000003167. PMID 33214495
- [Background] Gillespie A, Fink EL, Traino HM, Uversky A, Bass SB, Greener J, Hunt J, Browne T, Hammer H, Reese PP, Obradovic Z. Hemodialysis Clinic Social Networks, Sex Differences, and Renal Transplantation. Am J Transplant. 2017 Sep;17(9):2400-2409. doi: 10.1111/ajt.14273. Epub 2017 Apr 21. PMID 28316126
- [Background] Urbanski M, Browne T, Ghanta M, Constantinescu S, Gillespie A, Hammer H, Traino H. Transplant Professionals' Perceptions of Long-Term Care Residents' Candidacy for Kidney Transplantation. Prog Transplant. 2017 Jun;27(2):146-151. doi: 10.1177/1526924817699968. Epub 2017 Mar 22. PMID 28617165
- [Background] Gillespie A, Fink EL, Gardiner HM, Gadegbeku CA, Reese PP, Obradovic Z. Does Whom Patients Sit Next to during Hemodialysis Affect Whether They Request a Living Donation? Kidney360. 2021 Jan 15;2(3):507-518. doi: 10.34067/KID.0006682020. eCollection 2021 Mar 25. PMID 35369020
- [Background] Bass SB, Hollin IL, Kelly PJ, Alhajji M, D'Avanzo P, Maurer L, Gillespie A, Schatell D, Gardiner HM. Perceptions of live donor kidney transplantation using segmentation analysis and perceptual mapping to understand differences by self-reported health status in people on dialysis. Frontiers in Communication. 2022;6:785186. Doi: 10.3389/fcomm.2021.785186
- [Background] Mead EL, Doorenbos AZ, Javid SH, Haozous EA, Alvord LA, Flum DR, Morris AM. Shared decision-making for cancer care among racial and ethnic minorities: a systematic review. Am J Public Health. 2013 Dec;103(12):e15-29. doi: 10.2105/AJPH.2013.301631. Epub 2013 Oct 17. PMID 24134353
- [Background] Scientific Registry of Transplant Recipients. Program Specific Reports. Saint Barnabas Medical Center. https://www.srtr.org/document/pdf?fileName=\012022_release\pdfPSR\NJSBTX1KI202111PNEW.pdf. Accessed February 1, 2022
- [Background] Scientific Registry of Transplant Recipients. Program Specific Reports. Temple University Hospital. https://www.srtr.org/document/pdf?fileName=\012022_release\pdfPSR\PATUTX1KI202111PNEW.pdf. Accessed February 1, 2022.
- [Background] Creswell JW, Plano Clark VL. Designing and conducting mixed methods research. Thousand Oaks, CA: Sage; 2006
- [Background] Creswell JW, Plano Clark VL. Designing and conducting mixed methods research (3rd ed.). Thousand Oaks, CA: Sage; 2017
- [Background] Creswell JW, Fetters MD, Ivankova NV. Designing a mixed methods study in primary care. Ann Fam Med. 2004 Jan-Feb;2(1):7-12. doi: 10.1370/afm.104. PMID 15053277
- [Background] Watzlawick P, Bavelas JB, Jackson DD. Pragmatics of human communication: a study of interactional patterns, pathologies, and paradoxes. New York, NY: W. W. Norton & Company, Inc.; 1967.
- [Background] Burgoon JK, Hale JL. The fundamental topoi of relational communication. Communication Monographs. 1984;51(3):193. https://doi.org/10.1080/03637758409390195
- [Background] Andersen PA, Guerrero LK, Buller DB, Jorgensen PF. An empirical comparison of three theories of nonverbal immediacy exchange. Human Communication Research 1998;24(4):501-35. https://doi.org/10.1111/j.1468-2958.1998.tb00429.x
- [Background] Kiesler DJ, Auerbach SM. Integrating measurement of control and affiliation in studies of physician-patient interaction: the interpersonal circumplex. Soc Sci Med. 2003 Nov;57(9):1707-22. doi: 10.1016/s0277-9536(02)00558-0. PMID 12948579
- [Background] Roter D, Larson S. The Roter interaction analysis system (RIAS): utility and flexibility for analysis of medical interactions. Patient Educ Couns. 2002 Apr;46(4):243-51. doi: 10.1016/s0738-3991(02)00012-5. PMID 11932123
- [Background] Ford S, Hall A, Ratcliffe D, Fallowfield L. The Medical Interaction Process System (MIPS): an instrument for analysing interviews of oncologists and patients with cancer. Soc Sci Med. 2000 Feb;50(4):553-66. doi: 10.1016/s0277-9536(99)00308-1. PMID 10641807
- [Background] Siminoff LA, Step MM. A comprehensive observational coding scheme for analyzing instrumental, affective, and relational communication in health care contexts. J Health Commun. 2011 Feb;16(2):178-97. doi: 10.1080/10810730.2010.535109. PMID 21213170
- [Background] Step MM, Rose JH, Albert JM, Cheruvu VK, Siminoff LA. Modeling patient-centered communication: oncologist relational communication and patient communication involvement in breast cancer adjuvant therapy decision-making. Patient Educ Couns. 2009 Dec;77(3):369-78. doi: 10.1016/j.pec.2009.09.010. Epub 2009 Oct 6. PMID 19811883
- [Background] Step MM, Siminoff LA, Rose JH. Differences in oncologist communication across age groups and contributions to adjuvant decision outcomes. J Am Geriatr Soc. 2009 Nov;57 Suppl 2:S279-82. doi: 10.1111/j.1532-5415.2009.02512.x. PMID 20122030
- [Background] Stothers L, Gourlay WA, Liu L. Attitudes and predictive factors for live kidney donation: a comparison of live kidney donors versus nondonors. Kidney Int. 2005 Mar;67(3):1105-11. doi: 10.1111/j.1523-1755.2005.00176.x. PMID 15698451
- [Background] Bandura A. Guide for constructing self-efficacy scales. In: F Pajares and TC Urdan (Eds.). Self-Efficacy Beliefs of Adolescents, pp. 307-337. Greenwich, CT: Information Age Publishing; 2006
- [Background] Waterman AD, Robbins ML, Paiva AL, Peipert JD, Davis LA, Hyland SS, Schenk EA, Baldwin KA, Amoyal NR. Measuring kidney patients' motivation to pursue living donor kidney transplant: development of stage of change, decisional balance and self-efficacy measures. J Health Psychol. 2015 Feb;20(2):210-21. doi: 10.1177/1359105313501707. Epub 2013 Oct 22. PMID 24155194
- [Background] Pradel FG, Suwannaprom P, Mullins CD, Sadler J, Bartlett ST. Haemodialysis patients' readiness to pursue live donor kidney transplantation. Nephrol Dial Transplant. 2009 Apr;24(4):1298-305. doi: 10.1093/ndt/gfn733. Epub 2009 Jan 7. PMID 19131353
- [Background] Rodrigue JR, Cornell DL, Kaplan B, Howard RJ. Patients' willingness to talk to others about living kidney donation. Prog Transplant. 2008 Mar;18(1):25-31. doi: 10.1177/152692480801800107. PMID 18429579
- [Background] Barnieh L, McLaughlin K, Manns B, Klarenbach S, Yilmaz S, Hemmelgarn B; Alberta Kidney Disease Network. Development of a survey to identify barriers to living donation in kidney transplant candidates. Prog Transplant. 2009 Dec;19(4):304-11. doi: 10.1177/152692480901900404. PMID 20050452
- [Background] Reese PP, Shea JA, Berns JS, Simon MK, Joffe MM, Bloom RD, Feldman HI. Recruitment of live donors by candidates for kidney transplantation. Clin J Am Soc Nephrol. 2008 Jul;3(4):1152-9. doi: 10.2215/CJN.03660807. Epub 2008 Apr 2. PMID 18385392
- [Background] LaVeist TA, Nickerson KJ, Bowie JV. Attitudes about racism, medical mistrust, and satisfaction with care among African American and white cardiac patients. Med Care Res Rev. 2000;57 Suppl 1:146-61. doi: 10.1177/1077558700057001S07. PMID 11092161
- [Background] Wallace LS, Rogers ES, Roskos SE, Holiday DB, Weiss BD. Brief report: screening items to identify patients with limited health literacy skills. J Gen Intern Med. 2006 Aug;21(8):874-7. doi: 10.1111/j.1525-1497.2006.00532.x. PMID 16881950
- [Background] Morgan JC, Golden SD, Noar SM, Ribisl KM, Southwell BG, Jeong M, Hall MG, Brewer NT. Conversations about pictorial cigarette pack warnings: Theoretical mechanisms of influence. Soc Sci Med. 2018 Dec;218:45-51. doi: 10.1016/j.socscimed.2018.09.063. Epub 2018 Oct 3. PMID 30340152
- [Background] Borland R, Yong HH, Wilson N, Fong GT, Hammond D, Cummings KM, Hosking W, McNeill A. How reactions to cigarette packet health warnings influence quitting: findings from the ITC Four-Country survey. Addiction. 2009 Apr;104(4):669-75. doi: 10.1111/j.1360-0443.2009.02508.x. Epub 2009 Feb 10. PMID 19215595
- [Background] Spitzberg BH, Cupach WR. Interpersonal communication competence. Beverly Hills, CA: Sage; 1984
- [Background] Hargie O. Handbook of communication skills. New York: Routledge; 200
- [Background] Brown RF, Bylund CL. Communication skills training: describing a new conceptual model. Acad Med. 2008 Jan;83(1):37-44. doi: 10.1097/ACM.0b013e31815c631e. PMID 18162748
- [Background] Bos-van den Hoek DW, Visser LNC, Brown RF, Smets EMA, Henselmans I. Communication skills training for healthcare professionals in oncology over the past decade: a systematic review of reviews. Curr Opin Support Palliat Care. 2019 Mar;13(1):33-45. doi: 10.1097/SPC.0000000000000409. PMID 30562180
- [Background] Stiefel F, de Vries M, Bourquin C. Core components of Communication Skills Training in oncology: A synthesis of the literature contrasted with consensual recommendations. Eur J Cancer Care (Engl). 2018 Jul;27(4):e12859. doi: 10.1111/ecc.12859. Epub 2018 Jun 5. PMID 29873149
- [Background] Smith MB, Macieira TGR, Bumbach MD, Garbutt SJ, Citty SW, Stephen A, Ansell M, Glover TL, Keenan G. The Use of Simulation to Teach Nursing Students and Clinicians Palliative Care and End-of-Life Communication: A Systematic Review. Am J Hosp Palliat Care. 2018 Aug;35(8):1140-1154. doi: 10.1177/1049909118761386. Epub 2018 Mar 8. PMID 29514480
- [Background] Banerjee SC, Manna R, Coyle N, Penn S, Gallegos TE, Zaider T, Krueger CA, Bialer PA, Bylund CL, Parker PA. The implementation and evaluation of a communication skills training program for oncology nurses. Transl Behav Med. 2017 Sep;7(3):615-623. doi: 10.1007/s13142-017-0473-5. PMID 28211000
- [Background] Lubrano di Ciccone B, Brown RF, Gueguen JA, Bylund CL, Kissane DW. Interviewing patients using interpreters in an oncology setting: initial evaluation of a communication skills module. Ann Oncol. 2010 Jan;21(1):27-32. doi: 10.1093/annonc/mdp289. Epub 2009 Jul 21. PMID 19622593
- [Background] Pehrson C, Banerjee SC, Manna R, Shen MJ, Hammonds S, Coyle N, Krueger CA, Maloney E, Zaider T, Bylund CL. Responding empathically to patients: Development, implementation, and evaluation of a communication skills training module for oncology nurses. Patient Educ Couns. 2016 Apr;99(4):610-616. doi: 10.1016/j.pec.2015.11.021. Epub 2015 Nov 24. PMID 26686992
- [Background] McCambridge J, Witton J, Elbourne DR. Systematic review of the Hawthorne effect: new concepts are needed to study research participation effects. J Clin Epidemiol. 2014 Mar;67(3):267-77. doi: 10.1016/j.jclinepi.2013.08.015. Epub 2013 Nov 22. PMID 24275499
- [Background] Sedgwick P, Greenwood N. Understanding the Hawthorne effect. BMJ. 2015 Sep 4;351:h4672. doi: 10.1136/bmj.h4672. No abstract available. PMID 26341898
- [Background] Syed M, Nelson SC. Guidelines for establishing reliability when coding narrative data. Emerging Adulthood. 2015;3(6):375-87. DOI: 10.1177/2167696815587648
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] U.S. Department of Health and Human Services. Advancing American Kidney Health. 2019. https://aspe.hhs.gov/system/files/pdf/262046/AdvancingAmericanKidneyHealth.pdf. Accessed February 1, 2022
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343